CLINICAL TRIAL: NCT02670603
Title: A Prospective Randomized Controlled Trial of Evonail® Solution for Prevention or Treatment of Onycholysis in Breast Cancer Patients Who Received Neoadjuvant/Adjuvant Docetaxel Chemotherapy
Brief Title: A Trial of Evonail® Solution for Prevention or Treatment of Onycholysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yeon Hee Park, MD,Ph.D, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2015-04-018-002
Record Dates: First submitted 2016-01-28; First posted 2016-02-02 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer; Docetaxel Chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This study is open-labeled study. But outcome would be assessed the statistician who did not involve this study with blind data.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Experimental arm (Experimental): In experimental arm, each patient painted EVONAIL® solution on nails and periungual areas once a day till developing onycholysis grade 2 or more.
  Interventions: Drug: EVONAIL® solution
- Control arm (Other): In control arm, each patient painted EVONAIL® solution on nails and periungual area twice a day after developing onycholysis grade 2.
  This study design allowed cross-over. Therefore, this control arm would give EVONAIL® solution after developing onlycholysis grade 2 in spite of control arm.
  Interventions: Drug: EVONAIL® solution

INTERVENTIONS:
Drug: EVONAIL® solution
  Other Names: Hydrating Nail Solution

SUMMARY:
This study is a prospective randomized controlled study of EVONAIL® solution for prevention or treatment of onycholysis in patients with breast cancer receiving docetaxel chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with breast cancer receiving adjuvant/neoadjuvant docetaxel chemotherapy

Exclusion Criteria:

* Patients with breast cancer receiving palliative docetaxel chemotherapy
* Patients having onycholysis before docetaxel treatment

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
The incidence of onycholysis Gr 2 or more | 12weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JY, Ok ON, Seo JJ, Lee SH, Ahn JS, Im YH, Park YH. A prospective randomized controlled trial of hydrating nail solution for prevention or treatment of onycholysis in breast cancer patients who received neoadjuvant/adjuvant docetaxel chemotherapy. Breast Cancer Res Treat. 2017 Aug;164(3):617-625. doi: 10.1007/s10549-017-4268-7. Epub 2017 May 9. PMID 28488142